CLINICAL TRIAL: NCT02445638
Title: HDL Lipidomic, Proteomic and Functional Changes in Response to Whole Egg Consumption in Overweight and Obese Women
Brief Title: HDL Lipidomic, Proteomic and Functional Changes in Women After Eating Eggs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 693261
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole egg (Active Comparator): Subjects will be provided with a daily breakfast meal containing the equivalent of 2 whole eggs for 4 weeks.
  Interventions: Other: Whole egg
- Yolk-free egg (Placebo Comparator): Subjects will be provided with a daily breakfast meal containing the equivalent of 2 yolk-free eggs for 4 weeks.
  Interventions: Other: Yolk-free egg

INTERVENTIONS:
Other: Whole egg — Subjects will be provided with the equivalent of 2 whole eggs daily.
  Arms: Whole egg
Other: Yolk-free egg — Subjects will be provided with the equivalent of 2 yolk-free eggs daily.
  Arms: Yolk-free egg

SUMMARY:
The objective of this randomized, single blinded cross-over study is to investigate effects of daily egg versus yolk-free egg substitute consumption on High Density Lipoprotein (HDL) composition and function in a population of overweight and obese postmenopausal women.

DETAILED DESCRIPTION:
The investigators hypothesize that after 4 weeks of daily consumption of whole egg versus yolk-free egg will result in differences in the HDL composition and profile of lipids and proteins (lipidome and proteome), which will be associated with changes in HDL functionality. It is further hypothesized that it will be possible to discriminate between responders and non-responders to eggs in terms of increasing both apolipoprotein A-1 (ApoA-I) content in the plasma, corresponding with more protective HDL particles; and increasing HDL functionality (cholesterol efflux and anti-oxidant capacity).

Subjects will consume an egg free diet during study protocols, except for the egg meal provided by the study. The study is comprised of two 4-week feeding periods with a 4-week washout between testing periods. While on the study, subjects will consume the equivalent of two eggs for breakfast, either whole egg or yolk-free egg. Following a 2-week low-egg lead-in period, subjects will be randomly selected to start on either arm and cross over to the other arm after the 4-week washout period.

Measured results will be compared between the baseline and the 4-week end point for each arm. Additional comparisons may be made between 4-week endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45-70 years old
* Overweight or obese (BMI 25-35 kg/m2)
* Post-menopausal (confirmed by clinical hormone levels assessed at screening if within one year of last menses)
* Plasma HDL cholesterol greater than or equal to 50 mg/dL.

Exclusion Criteria:

* Documented chronic diseases including diabetes, thyroid disease, metabolic syndrome, cancer (active), or previous cardiovascular events
* Having 3 or more traits of Metabolic Syndrome
* Egg allergy or multiple food allergies or food intolerances that would significantly limit food intake
* Smoker
* Current consumption more than 1 alcoholic drink/ day
* Extreme dietary or exercise patterns
* Recent weight fluctuations (greater than 10% in the last six months)
* Anemia
* Taking prescription lipid medications or other supplements known to alter lipoprotein metabolism such as isoflavones, red yeast rice, or > 1 g of fish oil/day.
* Taking exogenous hormones (i.e. hormone replacement therapy)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline Apo A-1 concentration | 4 weeks
  The concentration of HDL Apo A-1 will be measured at baseline and after 4 weeks of whole egg, and after 4 weeks of yolk-free egg consumption, in randomized order.

SECONDARY OUTCOMES:
Change from baseline HDL function | 4 weeks
  Parameters of HDL functionality (i.e. cholesterol efflux and anti-oxidant function) will be measured at baseline and after 4 weeks of whole egg, and after 4 weeks of yolk-free egg consumption, in randomized order.
Change from baseline HDL composition | 4 weeks
  The lipidomic and proteomic profiles of HDL will be measured at baseline and after 4 weeks of whole egg and after 4 weeks of yolk-free egg consumption, in randomized order.

CONTACTS AND LOCATIONS:
Overall Officials: Francene Steinberg, PhD, RD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

REFERENCES:
- [Derived] Sawrey-Kubicek L, Zhu C, Bardagjy AS, Rhodes CH, Sacchi R, Randolph JM, Steinberg FM, Zivkovic AM. Whole egg consumption compared with yolk-free egg increases the cholesterol efflux capacity of high-density lipoproteins in overweight, postmenopausal women. Am J Clin Nutr. 2019 Sep 1;110(3):617-627. doi: 10.1093/ajcn/nqz088. PMID 31172172